CLINICAL TRIAL: NCT00712465
Title: A Phase I, Randomised, Open, Single-centre, Three-period Crossover Study to Evaluate the Effect of AZD1305 on the Pharmacokinetics of Digoxin After Repeated Oral Administration of AZD1305 and Digoxin to Young Healthy Male Volunteers
Brief Title: An Interaction Study With Digoxin and AZD1305
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmia and Lipids, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3190C00010; 2008-000577-37 (EudraCT No)
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; interaction; pharmacokinetic
MeSH Terms: conditions — Atrial Fibrillation | interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AZD1305 tablet
  Interventions: Drug: AZD1305
- 2 (Experimental): AZD1305 tablet + digoxin
  Interventions: Drug: AZD1305; Drug: Digoxin
- 3 (Active Comparator): Digoxin
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: AZD1305 — Extended Release tablet, repeated administration
  Arms: 1; 2
Drug: Digoxin — Tablet, repeated administration
  Arms: 2; 3

SUMMARY:
The primary purpose of this study is to learn more about how digoxin is handled by the body, i.e. absorption, distribution, metabolism and excretion, when administered alone and in combination with AZD1305. Secondary purposes are to learn more about how AZD1305 is handled by the body when administered alone and in combination with digoxin and to learn more about how AZD1305 and digoxin administered alone and in combination affect the body.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI=weight/height2) of 19 to 30 kg/m2

Exclusion Criteria:

* Potassium outside normal reference values
* ECG findings outside normal range

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables | During all dosing visits

SECONDARY OUTCOMES:
Adverse event, vital signs, ECG, physical examination and laboratory variables. | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Marianne Hartford, MD, PhD, Principal Investigator — AstraZeneca, Clinical Pharmacology Unit, Sahlgrenska University Hospital
Locations (1):
- Research Site, Gothenburg, Sweden